CLINICAL TRIAL: NCT04769024
Title: Evaluation of the Benefits of an Immersive Virtual Reality Intervention (LUMEEN) for Behavioral and Psychological Symptoms of Dementia in People Living in Residential Aged Care.
Brief Title: Virtual Reality Intervention for the Reduction of Behavioral and Psychological Symptoms of Dementia
Acronym: LUMEENCOMPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 69HCL20_1246
Record Dates: First submitted 2021-02-08; First posted 2021-02-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Alzheimer's Disease; Neurocognitive Disorders
Keywords: BPSD; Dementia; Apathy; virtual reality; Alzheimer's disease; Neurocognitive Disorders
MeSH Terms: conditions — Dementia; Alzheimer Disease; Neurocognitive Disorders; Lethargy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUMEEN intervention (Active Comparator): Participants in the LUMEEN intervention group will participate in the 12 LUMEEN Virtual Reality sessions of 45 minutes taking place twice a week for 6 weeks, in groups of 6 participants. The content of these sessions is described in the Intervention Description part of this document.
  Interventions: Device: LUMEEN Virtual Reality sessions
- USUAL activities (Sham Comparator): Participants in the control group will participate in the 12 Control/non-digital stimulation sessions of 45 minutes taking place twice a week for 6 weeks, in groups of 6 participants instead of the LUMEEN Virtual Reality sessions. The content of these sessions is described in the Intervention Description part of this document.
  Interventions: Behavioral: Control/non-digital stimulation sessions

INTERVENTIONS:
Device: LUMEEN Virtual Reality sessions — It will consist in carrying out 12 virtual reality sessions in groups of 6 participants, at a rate of 2 per week for approximately 6 weeks, using the LUMEEN "EVASION" module. Each session lasts approximately 45 minutes. This module allows the simultaneous broadcasting in virtual reality headsets of 360° videos accompanied by music about different themes: nature, animals, travel, art and live performance.
  The course of an EVASION session is as follows:
  1. The participants are seated in armchairs in an open environment and sufficiently spaced so that they can move their arms without bumping into each other.
  2. The facilitator announces the immersion theme of the session
  3. Participants are equipped with virtual reality head-mounted displays.
  4. Participants watch the content.
  5. The head-mounted displays are removed.
  6. A group discussion encouraging participants to share their feelings and what they have learned from the immersion is conducted by the facilitator.
  Arms: LUMEEN intervention
Behavioral: Control/non-digital stimulation sessions — It will consist in non-digital stimulation (sensory, social, cognitive, creative) group sessions offering various typical pen-and-paper activities for this public which mainly stimulate language, immediate memory, semantic memory, and visual recognition (e.g., definitions, games of 7 differences, reconstruction of proverbs, quizzes…). A set of activities with instructions will be provided to the investigating centres but the choice of activities in each session will be left to the facilitator's decision in order to adapt the sessions to the participants' desires and abilities, as is usually done in such stimulation groups. The sessions will last 45 minutes and will be offered twice a week for 6 weeks by a facilitator or a caregiver with group care training. The sessions will be organized in groups of 6 participants to match the group size of the intervention groups.
  Arms: USUAL activities

SUMMARY:
Alzheimer's disease and related disorders (AD2) are characterised by cognitive changes and Behavioural and Psychological Symptoms of Dementia (BPSD). According to the French National Authority for Health (2009), Non-Pharmacological Interventions (N PhIs) are to be favo red in the treatment of BPSD. A few NPhIs have already shown their effectiveness in the management of these symptoms, such as music therapy or multi-sensory stimulation, but these techniques require trained staff and/or adapted premises. Over the past decade, innovative techniques have emerged in the field of NPhIs. Virtual Reality (VR) is one of them. Amongst the VR tools, the LUMEEN technology offers a suitable mediation tool for older adults with disabilities which allows to show immersive experiences in calm landscapes known to bring a feeling of well-being (beach, mountain, dolphins, classical music concert, animals in nature, etc.).

The main objective of this study is to evaluate the effect of the LUMEEN Evasion module on the occurrence of BPSD in older adults living in residential aged care.

Participants will be recruited in nursing homes and randomly assigned to the LUMEEN intervention group or the control group. Participants in the LUMEEN intervention group will attend 12 LUMEEN group session s in which they will be immersed for a few minutes in a selection of landscapes or scenes using virtual reality head-mounted displays and will then have a group discussion about the immersive experience they watched during the session. Participants in the control group will attend 12 non-digital (sensory, social, cognitive, creative) stimulation group sessions in which they will carry out typical pen-and-paper activities for this public which mainly stimulate language, immediate memory, semantic memory, and visual recognition (e.g., definitions, games of 7 differences, reconstruction of proverbs, quizzes…).

The BPSD will be evaluated by the healthcare team before the start of the intervention and after the 12 sessions in both arms of the study (LUMEEN intervention and control) using the Neuropsychiatric Inventory filled out by the nursing staff (NPI). LUMEEN sessions are expected to reduce BPSD (especially apathy) more than control sessions. Thus, participants in the LUMEEN intervention group should have a greater difference between baseline and post-intervention NPI scores than the participants in the control group (in the direction of a reduction of the symptoms in the post-intervention evaluation).

Secondary outcomes will also be measured focusing on apathy, well-being and social interactions. First of all, apathy will be evaluated thanks to the Apathy Inventory - Clinician before and after the interventions in both groups. Then, the state of well-being of the participant will be evaluated thanks to the EVIBE scale completed before and after each session. In addition, social interaction behaviors will be rated using the Social Behaviour Resident Index (SOBRI), collected through a 4-minutes participant observation during each session by an external observer.

LUMEEN sessions are expected to improve these three outcomes more than control sessions. Differences are expected to be observed between the two groups : a) apathy should be lower after the sessions than before and the pre-post-intervention difference should be larger in the LUMEEN intervention group than in the control group; b) well-being should be (in average) higher after the sessions than before and the pre-post-intervention difference should be larger in the LUMEEN intervention group than in the control group ; and c) there should be, on average, more social interactions behaviours during the LUMEEN sessions than during the control sessions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have to present a NPI score of 9 or more on at least one of the following items : apathy, agitation, anxiety, depression, aberrant motor behavior.
* The behavioural disorders do not prevent the participation in a session.
* For participants able to give consent:

  * Written informed consent to participate in the study
  * Informed consent of the participant in the presence of his/her curator for participant under curatorship.
* For participants who are not able to receive information and to give consent:

  * Written informed consent of the legal representative (tutor) for participants under tutelage.
  * Signature of a relative (family member and/or trusted person) of the participant
* The participant has to be affiliated to a social security scheme.

Exclusion Criteria :

* Unstable pathology whose nature may interfere with the assessment variables:

  * Neurological disorder of infectious origin
  * Psychiatric disorder
  * Substance abuse
* Severe uncompensated sensory deficit
* History of epilepsy
* Pacemaker or severe and/or uncontrolled heart disease (at the discretion of the investigator)
* Visual hallucinations
* Burns and sores on the upper face or scalp
* Unable to express their consent, without a trusted person (family or close friend) and not legally protected

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Differences in Neuropsychiatric Inventory filled out by the nursing staff (NPI) score between before and after the intervention | 12 weeks
  The NPI is used to assess the behavioural and psychological symptoms often associated with neurocognitive disorders and dementia. We will compare both groups (LUMEEN intervention and Control) on the differences in NPI scores collected before and after the intervention.

SECONDARY OUTCOMES:
Differences between the mean EVIBE scores before the sessions and the mean EVIBE scores after the sessions compared between the two groups (Lumeen intervention and control). | 12 weeks
  It is a visual analogue scale to report on one's own state of well-being. In response to the question "How do you feel right now?", the participant estimates his/her sense of well-being based on pictograms representing simple facial expressions. The participant's position according to the pictograms correspond to a numerical value from 1 to 5. "1" corresponds to the lowest feeling of well-being and "5" to the highest feeling of well-being. The difference of means between scores observed before and after the intervention will be compared between groups.
Differences between scores on the Apathy Inventory - Clinician (AI-Clinician) completed before and after the 12 intervention sessions, compared between the LUMEEN intervention group and the control group. | 12 weeks
  The Apathy Inventory - Clinician collects information on the presence of apathy according to three dimensions: emotional blunting, loss of initiative, loss of interest. Each dimension is assessed by a clinician according to its frequency (1: sometimes, 2: fairly often, 3: frequently, 4; very frequently) and severity (1: mild, 2: moderate, 3: severe). The score for each dimension is calculated by multiplying the frequency by the severity, resulting in a maximum score of 12. The total score of the AI-Clinician is obtained by adding the scores of the 3 dimensions, obtaining a maximum score of 36.
Mean of the Social Behaviour Resident Index (SOBRI) scores completed during each session, compared between LUMEEN intervention and control groups | 12 weeks
  The SOBRI is used to observe and objectify social interaction behaviours. It consists of two components: social interactions between residents (10 interaction types) and social interactions between residents and staff (6 interaction types). Social interactions are analysed in terms of presence or absence

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - EHPAD du Centre Hospitalier du Pays de Craponne Sur Arzon, Craponne-sur-Arzon
  - EHPAD du Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - EHPAD Saint-Joseph, Le Puy-en-Velay
  - EHPAD Maison Saint-François d'Assise Lyon, Lyon
  - EHPAD Korian Saison Dorée, Lyon
  - EHPAD Korian Les Aurélias, Pollionnay

IPD SHARING:
Plan to Share IPD: Undecided